CLINICAL TRIAL: NCT03571347
Title: Refugee Emergency: DEFining and Implementing Novel Evidence-based Psychosocial Interventions
Brief Title: Self Help Plus for Asylum Seekers and Refugees in Europe
Acronym: REDEFINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: World Health Organization (Other); VU University of Amsterdam (Other); University of Vienna (Other); University of Ulm (Other); The International Federation of Red Cross and Red Crescent Societies (Other); University of Turku (Other); University of Liverpool (Other); University of York (Other)
Responsible Party: Principal Investigator, Marianna Purgato, Principal Investigator, PhD, Clinical researcher, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 779255
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Stress, Psychological
Keywords: distress; post-traumatic stress disorder; prevention; asylum seekers; refugees; Self Help Plus; Europe
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: RE-DEFINE is a prospective, multicentre, randomized, parallel-group trial that will follow study participants over a period of 12-months. Asylum seekers and refugees with psychological distress, but without a mental disorder according to the MINI International Neuropsychiatric Interview (M.I.N.I.) for DSM-V and ICD-10, will be randomly assigned to the Self Help Plus intervention or to enhanced treatment as usual (ETAU).
Who Masked: Outcomes Assessor
Masking Description: Participants, facilitators, and research staff involved in the screening and baseline assessment will not be blind to the interventions provided during the trial. Outcomes assessors will be kept blind to the study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Help Plus (Experimental): SH+ programme has been developed by WHO and collaborators working in the humanitarian field, with expertise in global mental health and psychosocial interventions. SH+ programme consists of a pre-recorded audio course, complemented with bibliotherapy, and thanks to this format not requiring much time from experts for implementation. SH+ consists of 5 sessions.
  Interventions: Behavioral: Self Help Plus
- Enhanced Treatment As Usual (Other): Control arm participants will receive routine social support and/or care according to ordinary practice and following local regulations. Additionally, they will receive baseline and follow-up assessments according to the study schedule, and information about freely available mental health services, social services and community networks providing support to asylum seekers and refugees, and NGOs' contact details.
  Interventions: Other: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Self Help Plus — 5-session psychosocial intervention
  Arms: Self Help Plus
Other: Enhanced Treatment As Usual — Routine social support and/or care, and information about freely available mental health services, social services, NGOs, and community networks providing support to asylum seekers and refugees
  Arms: Enhanced Treatment As Usual

SUMMARY:
Background The flow of asylum seekers and refugees moving to European and bordering countries has progressively increased in the last years. This population is exposed to physical and mental challenges before and during displacement, and suffer continuing hardships after arrival in a High-Income Country. As a consequence, asylum seekers and refugees are extremely vulnerable to some common mental health conditions, i.e., post-traumatic stress disorder, anxiety, depression and other forms of disabling psychological distress. The World Health Organization has developed a new 5-session self-help intervention called Self-Help Plus (SH+) for managing stress and coping with adversity. SH+ has been evaluated in RCTs in low- and middle-income countries, however, there is no rigorous evidence on its cost-effectiveness in preventing the onset of mental disorders in HIC.

Objectives To evaluate the effectiveness and cost-effectiveness of the SH+ in asylum seekers and refugees with psychological distress resettled in six sites of five European countries (Italy, Austria, Germany, Finland, and two sites in the UK), as compared with enhanced treatment as usual (ETAU). The primary outcome is the reduction in the incidence of any mental disorders. Secondary outcomes are mental health symptoms, psychological functioning, well-being, drop-out rates, and economic outcomes.

Design This is a multicentre parallel-group randomized controlled trial, in which participants will have an equal probability (1:1) of being randomly allocated to the SH+ or the ETAU.

Methodology Asylum seekers and refugees who screen positive at the General Health Questionnaire (≥ 3) and without a formal diagnosis of any psychiatric disorders according to the M.I.N.I. International Neuropsychiatric Interview will enter the study. After random allocation they will receive the SH+ or the ETAU. Assessments will be performed by masked assessors immediately after intervention, at 6 months, and a 12 months after randomization.

Time frame The recruitment phase will last 12 months. After the screening, eligible participants will be assessed at baseline, post-intervention, and at 6- and 12-month follow-up. The SH+ delivery will be conducted in around 5 weeks.

Expected outcomes A reduction in the incidence of psychiatric diagnoses at 6-month follow-up, and a general improvement in mental health symptoms, psychological functioning, well-being, and economic outcomes at each assessment.

DETAILED DESCRIPTION:
Asylum seekers and refugees will be randomized to receive the SH+ intervention or Enhanced Treatment as Usual. The SH+ has been developed by WHO and collaborators working in the humanitarian field, with expertise in global mental health and psychosocial interventions. SH+ consists of a pre-recorded audio course, delivered by facilitators in a group setting and complemented with an illustrated self-help book. SH+ was designed to be relevant for large adversity-affected populations: it is transdiagnostic, easily adaptable to different cultures and languages, and both meaningful and safe for people with and without mental disorders. The format of SH+ is innovative in that it seeks to ensure that key intervention components are delivered as intended without the burden of extensive facilitator training. SH+ programme is based on acceptance and commitment therapy (ACT), a form of cognitive-behavioral therapy, with distinct features. SH+ programme has two components: a pre-recorded course and an illustrated self-help book. Pre-recorded audio material (culturally adapted) is delivered across five 2-hour sessions to groups of up to 30 people. The audio material imparts key information about stress management and guides participants through individual exercises and small group discussions. To augment the audio recordings, an illustrated self-help book reviews all essential content and concepts 19. Written manuals help briefly-trained, non-specialist facilitators to conduct the course using the pre-recorded audio. The SH+ intervention will be delivered by briefly-trained, non-specialist facilitators.

The control intervention will receive Enhanced Treatment as Usual.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above;
2. Able to speak and understand the target languages: Arabic, and/or Urdu, and/or Dari, and/or English;
3. Asylum seeker or refugee;
4. Presence of psychological distress, as shown by a score of 3 or more at the 12 item General Health Questionnaire (GHQ-12 ≥ 3);
5. Both oral and written informed consent to enter the study.

Exclusion Criteria:

1. Presence of any mental disorders according to DSM-V and ICD-10, as shown by a positive M.I.N.I.;
2. Acute medical conditions contraindicating study participation, based on clinical judgment of the health care professional with a clinical background who performs the screening;
3. Clinical evidence of imminent suicide risk or suicide risk scored as "moderate or high" (or a positive suicidality behaviour disorder) by the M.I.N.I. (section SUICIDALITY);
4. Clinical evidence that the decision-making capacity is impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Psychiatric diagnosis at 6-month follow-up | 6-month follow-up
  The primary outcome will be the number of participants with a current psychiatric diagnosis 6 at six-month follow-up, as measured by the M.I.N.I.

SECONDARY OUTCOMES:
Psychological distress | Post-intervention; 6-month and 12-month follow-ups
  Psychological distress will be measured through the General Health Questionnaire-12. The questionnaire asks whether the respondent has experienced a particular symptom or behaviour recently. Each item is rated on a four-point Likert scale (less than usual, no more than usual, rather more than usual, or much more than usual); and gives a total score of 36 or 12 based on the GHQ version and on the selected scoring methods.
Psychiatric diagnosis | Post-intervention; 6-month and 12-month follow-ups
  Number of participants with a current psychiatric diagnosis as measured by the M.I.N.I.
Functioning | Post-intervention; 6-month and 12-month follow-ups
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) is a generic assessment instrument assessing health and disability. It is used across all diseases, including mental, neurological and substance use disorders. It is simple to administer and applicable across cultures.
Depressive symptoms | Post-intervention; 6-month and 12-month follow-ups
  Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item instrument measuring the presence and severity of depression. Major depression is diagnosed if five or more of the nine depressive symptom criteria have been present at least "more than half the days" in the past two weeks, and one of the symptoms includes depressed mood or anhedonia.
Subjective wellbeing | Post-intervention; 6-month and 12-month follow-ups
  WHO-5 Wellbeing index. The WHO-5 Wellbeing Index is a 5-item questionnaire measuring current psychological wellbeing and quality of life, rather than psychopathology.
Self-defined psychosocial goals | Post-intervention; 6-month and 12-month follow-ups
  The Psychological Outcome Profiles instrument (PSYCHLOPS) consists of four questions. It contains three domains: problems (2 questions), function (1 question) and wellbeing (1 question).
Symptoms of Post traumatic stress disorder | Post-intervention; 6-month and 12-month follow-ups
  PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.
Health-related quality of life | 6-month and 12-month follow-ups
  The EuroQol-5Dimension-3 level version (EQ-5D-3L). The EQ-5D-3L is applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.
Cost-effectiveness | 6-month and 12-month follow-ups
  The Client Service Receipt Inventory, European version (CSSRI-EU): Client sociodemographic and service receipt inventory (adapted version with other socio- demographic characteristics). The CSSRI is a research tool developed for collecting information that describes in detail the types and level of services that comprise the care package of each study member.
Proportion of participants leaving the study early | This information will be collecfted at any time.
  Number of people leaving the study prematurely at any times, and reasons for discontinuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Verona, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Purgato M, Carswell K, Acarturk C, Au T, Akbai S, Anttila M, Baumgartner J, Bailey D, Biondi M, Bird M, Churchill R, Eskici S, Hansen LJ, Heron P, Ilkkursun Z, Kilian R, Koesters M, Lantta T, Nose M, Ostuzzi G, Papola D, Popa M, Sijbrandij M, Tarsitani L, Tedeschi F, Turrini G, Uygun E, Valimaki MA, Wancata J, White R, Zanini E, Cuijpers P, Barbui C, Van Ommeren M. Effectiveness and cost-effectiveness of Self-Help Plus (SH+) for preventing mental disorders in refugees and asylum seekers in Europe and Turkey: study protocols for two randomised controlled trials. BMJ Open. 2019 May 14;9(5):e030259. doi: 10.1136/bmjopen-2019-030259. PMID 31092670